CLINICAL TRIAL: NCT00001015
Title: A Multicenter Phase I Clinical Trial of Ribavirin in the Treatment of Patients With AIDS and Advanced AIDS Related Illnesses
Brief Title: A Study of Ribavirin in the Treatment of Patients With AIDS and AIDS-Related Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 034; 11010 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Ribavirin; T-Lymphocytes; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
To determine the maximum long-term dosage of ribavirin (RBV) that is safe and free of serious side effects in patients with AIDS or AIDS related illnesses. Also, to determine what effect different dosage levels have on biologic markers of efficacy, such as the amount of the AIDS virus (HIV) or number of T cells in the patient's blood.

RBV is a new drug capable of inhibiting the growth of the AIDS virus in the laboratory with little effect on normal human cells. In earlier tests of RBV in AIDS patients, the drug was well tolerated and safe, and this favorable result suggested that RBV should be more extensively studied in patients with AIDS and advanced AIDS related complex (ARC).

DETAILED DESCRIPTION:
RBV is a new drug capable of inhibiting the growth of the AIDS virus in the laboratory with little effect on normal human cells. In earlier tests of RBV in AIDS patients, the drug was well tolerated and safe, and this favorable result suggested that RBV should be more extensively studied in patients with AIDS and advanced AIDS related complex (ARC).

Patients are selected from three patient groups:

* Patients with AIDS, who have not taken zidovudine (AZT) within 30 days of entry into the study and who have not been discontinued from AZT because of intolerance.
* Patients with AIDS related diseases who have not taken AZT within 30 days of entry into the study, and who have not been discontinued from AZT because of intolerance.
* Patients with AIDS or AIDS related diseases who have had AZT intolerance that required cessation of therapy. This is an outpatient study; patients are seen weekly for the first 4 weeks, every other week through week 12, and then every 4 weeks for the duration of the 24 weeks of the treatment portion of the study. Patients from each of the three diagnostic groups are enrolled at each dose level. For the first 3 days after entry into the study, all patients receive the lowest dose of RBV every 6 hours. Subsequent dosages increase until the maximum tolerated dose (MTD) is reached. The MTD for a group is defined as the dose at which 4 or more of the 8 patients in the group develop toxicity which requires a change or discontinuation of the dosage.

Patients who experience significant toxicity may continue in the study at lower dose to determine the long-term tolerance.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Short-course therapy (7 days) with oral acyclovir.
* Short-course therapy (7 days) with ketoconazole.
* Topical medications.
* Aerosolized pentamidine for prophylactic purposes.

Concurrent Treatment:

Allowed:

* Blood transfusions for hemoglobin toxicity.

Patients must have two positive HIV p24 antigen tests with titers = or > 70 picograms at least 72 hours apart and within 1 month prior to entry, the last of which must be within 2 weeks of starting therapy.

Prior Medication:

Allowed:

* Zidovudine (AZT), without cessation of therapy required due to intolerance.
* AZT therapy must be discontinued at least 30 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Active opportunistic infection, symptomatic visceral Kaposi's sarcoma (KS) or progression of KS within the month prior to entry into the study, neoplasms other than KS, basal cell carcinoma of the skin, or in situ carcinoma of the cervix. Significant diarrhea, defined as = or > 3 liquid stools per day within the past week.

Concurrent Medication:

Excluded:

* Ongoing systemic therapy and/or prophylaxis for an AIDS-defining opportunistic infection.
* Antineoplastic therapy.
* Other experimental medications.
* Systemic chemoprophylaxis for Pneumocystis carinii pneumonia.
* Chronic (> 7 days) oral acyclovir therapy.

Concurrent Treatment:

Excluded:

* Blood transfusions unless they are for = or > grade 3 hemoglobin toxicity.

Patients with the following are excluded:

* Active opportunistic infection, symptomatic visceral Kaposi's sarcoma (KS) or progression of KS within the month prior to entry into the study, neoplasms other than KS, basal cell carcinoma of the skin, or in situ carcinoma of the cervix. Significant diarrhea, defined as = or > 3 liquid stools per day within the past week.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretroviral agents including zidovudine (AZT).
* Biologic modifiers.
* Systemic corticosteroids.

Prior Treatment:

Excluded within 2 months of study entry:

* Blood transfusion except for those who have taken zidovudine (AZT) who may not have received a transfusion within the previous month.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Study Completion 1990-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crumpacker C, Study Chair
Locations (5):
- United States (5):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Background] Crumpacker C, Pearlstein G, van der Horst C, Valentine F, Spector S, Mills J. A phase one increasing dose trial of oral ribavirin (RBV) in patients with AIDS and ARC. Int Conf AIDS. 1990 Jun 20-23;6(3):203 (abstract no SB468)
- [Background] Crumpacker C, Cotton D, Pearlstein G, Valentine F, Mills J, Spector S. Ribavirin dose escalating phase 1 trial in patients with AIDS and ARC. Int Conf AIDS. 1989 Jun 4-9;5:336 (abstract no TBP296)